CLINICAL TRIAL: NCT00590265
Title: Light-Therapy in the Treatment of the Acute Phase of the Bipolar Type II Depression: Double-Blind, Placebo-Controlled Study to Establish Efficacy and Safety
Brief Title: Light-Therapy in the Treatment of the Acute Phase of the Bipolar Type II Depression
Acronym: BPII-DEP-LT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Douglas Mental Health University Institute (Other)
Collaborators: National Alliance for Research on Schizophrenia and Depression (Other)
Responsible Party: Principal Investigator, Serge Beaulieu, Serge Beaulieu, Douglas Mental Health University Institute
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NARSAD-9818
Record Dates: First submitted 2007-12-26; First posted 2008-01-10 (Estimated); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Bipolar Type II Disorder; Depression, Bipolar
Keywords: bipolar type II disorder; depression; remission; light-therapy; efficacy; safety
MeSH Terms: conditions — Bipolar Disorder; Depression | interventions — Ultraviolet Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental)
  Interventions: Device: Northern Light Technology (SADelite lamp) bright light-therapy
- 2 (Placebo Comparator)
  Interventions: Device: Northern Light Technology (SADelite lamp) Dim light-therapy

INTERVENTIONS:
Device: Northern Light Technology (SADelite lamp) bright light-therapy — 10 000 lux for 30 minutes
  Other Names: Northern Light Technology (SADelite lamp) with two 36W bulbs
  Arms: 1
Device: Northern Light Technology (SADelite lamp) Dim light-therapy — <100 lux for 30 minutes
  Other Names: Northern Light Technology (SADelite lamp) with two 18W bulbs + red filter (Medium Red 27 High Temperature treated, LEE Filters, Y = 3.64%)
  Arms: 2

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of light therapy for the treatment of bipolar type II patients relapsing into a depressive phase during autumn or winter.

DETAILED DESCRIPTION:
Bipolar type II depression is a very frequent condition for which we still have a significant lack of acute treatments. There is now consistent evidence that light-therapy treatment produced a significant decrease of depressive symptoms for seasonal and non-seasonal unipolar depression. But there are no long-term studies of light therapy for the treatment of non-seasonal unipolar depression. It is also important to note that many of these studies involved co-therapy with antidepressant drugs or sleep-deprivation, making the interpretation of the results even more difficult.

Therefore, we propose to study the efficacy and safety of light therapy for the treatment of bipolar type II patients relapsing into a depressive phase during the period of September to mid-March. This will be a double-blind randomized placebo-controlled study. Bipolar II out-patients will be recruited from our bipolar disorders program and from our 5 general psychiatry out-patient clinics. We will recruit bipolar type II patients facing a depressive phase and after they give their informed consent and we had verified they meet all inclusion and exclusion criteria, they will be randomized blindly to Bright-light (10 000 lux) vs Dim-light placebo (100 lux) therapies. Both, patient and investigator/rater will be blind to the type of light treatment assigned to the patient. The light therapy will take place during 30 minutes daily in the morning AFTER the usual awakening time of the patient in order to avoid even partial sleep deprivation which would confound the results if we were to observe a greater switch rate into mania or hypomania.

Reasons for study termination can be serious side-effects, development of suicidal ideations or hypomanic/manic symptoms, patient's own decision, or any other of the exclusion criteria being fulfilled during the course of the study.

Depressive and manic/hypomanic symptoms, quality of life, sleep quality and side-effects will be assessed at baseline and during the study. Biological parameters will also be measured along the study. We think that this study will allow us to determine the efficacy and safety of a 5 weeks bright light therapy for Bipolar type II depression and provide open label data as to the long term benefits of this treatment if prolonged over 5 weeks during the "dark" months of the year.

ELIGIBILITY:
Inclusion Criteria:

* Bipolar type II disorder, depressive phase meeting DSM-IV criteria as per the SCID interview
* Hamilton Depression Rating Scale 21 items (HAMD-21) ≥ 17 and a Montgomery Asberg rating Scale (MADRS) ≥ 15 for at least 2 weeks and the episode has begun during the month of september or a later month
* Able to give their consent and willingness to participate to the study

Exclusion Criteria:

* Other psychiatric condition, organic brain disorder, unstable and/or untreated medical condition such as hypothyroidism, diabetes, cardiac condition, hypertension
* Deficit in vitamin B12 or folate
* Sub-syndromic hypomania symptoms as per a Young Mania Rating Scale (YMRS) score ≥ 4
* History of manic or hypomanic switch when exposed to bright light or during prolonged exposure to the sun during previous depressive phases
* Pregnancy or absence of a contraceptive treatment
* History of light-induced migraine or epilepsy
* Marked suicidal ideation
* Retinal blindness or severe cataract
* Glaucoma, retinal diseases of the eye
* Alcohol or drug abuse
* Known skin sensitivity to sunlight, especially in patients receiving photosensitizing drugs such as lithium or phenothiazines
* Past history of light therapy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2008-01; Primary Completion 2025-06 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
the response rate as defined by a 50% improvement of the depressive symptoms score on the MADRS scale | 5 and 45 weeks

SECONDARY OUTCOMES:
the remission rate (MADRS scale ≤ 8 ) | 5 and 45 weeks
the relapse rate into depression or hypomania | 5 and 45 weeks
the sleep quality as per PSQI scale | 5 and 45 weeks
the quality of life as per SF-36 and Q-LES-Q SF scales | 5 and 45 weeks
the incidence of side-effects as per the UKU scale | 5 and 45 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Serge Beaulieu, Ph.D., Principal Investigator — McGill University
Locations (1):
- Douglas Mental Health University Institute, Montreal, Quebec, Canada

REFERENCES:
- [Background] Bauer MS, Shea N, McBride L, Gavin C. Predictors of service utilization in veterans with bipolar disorder: a prospective study. J Affect Disord. 1997 Jul;44(2-3):159-68. doi: 10.1016/s0165-0327(97)00046-3. PMID 9241576
- [Background] Devilly GJ, Borkovec TD. Psychometric properties of the credibility/expectancy questionnaire. J Behav Ther Exp Psychiatry. 2000 Jun;31(2):73-86. doi: 10.1016/s0005-7916(00)00012-4. PMID 11132119
- [Background] Golden RN, Gaynes BN, Ekstrom RD, Hamer RM, Jacobsen FM, Suppes T, Wisner KL, Nemeroff CB. The efficacy of light therapy in the treatment of mood disorders: a review and meta-analysis of the evidence. Am J Psychiatry. 2005 Apr;162(4):656-62. doi: 10.1176/appi.ajp.162.4.656. PMID 15800134
- [Background] Kripke DF, mullaney DJ, Gillin JC, et al. Phototherapy of non-seasonal depression. In: Shagass C, Josiassen RC, Bridger WH, et al., eds. Biological Psychiatry. New York: Elsevier Science Publishing Co.; 1986:993-995
- [Background] Kripke DF. Light treatment for nonseasonal depression: speed, efficacy, and combined treatment. J Affect Disord. 1998 May;49(2):109-17. doi: 10.1016/s0165-0327(98)00005-6. PMID 9609674
- [Background] Lam RW, Levitt AJ, Kraus RP, et al. Management issues. In: ed.R.Lam and A.Levitt, ed. Canadian Consensus Guidelines for the Treatment of Seasonal Affective Disorder Clinical & Academic Publishing; 1999:96-114
- [Background] Magnusson A, Partonen T. The diagnosis, symptomatology, and epidemiology of seasonal affective disorder. CNS Spectr. 2005 Aug;10(8):625-34; quiz 1-14. doi: 10.1017/s1092852900019593. PMID 16041294
- [Background] Martiny K, Lunde M, Unden M, Dam H, Bech P. The lack of sustained effect of bright light, after discontinuation, in non-seasonal major depression. Psychol Med. 2006 Sep;36(9):1247-52. doi: 10.1017/S0033291706008105. Epub 2006 Jun 7. PMID 16756691
- [Background] Schwitzer J, Neudorfer C, Blecha HG, Fleischhacker WW. Mania as a side effect of phototherapy. Biol Psychiatry. 1990 Sep 15;28(6):532-4. doi: 10.1016/0006-3223(90)90489-o. No abstract available. PMID 2132555
- [Background] Stout RL, Wirtz PW, Carbonari JP, Del Boca FK. Ensuring balanced distribution of prognostic factors in treatment outcome research. J Stud Alcohol Suppl. 1994 Dec;12:70-5. doi: 10.15288/jsas.1994.s12.70. PMID 7723001
- [Background] Tuunainen A, Kripke DF, Endo T. Light therapy for non-seasonal depression. Cochrane Database Syst Rev. 2004;2004(2):CD004050. doi: 10.1002/14651858.CD004050.pub2. PMID 15106233
- [Background] Wirz-Justice A, Benedetti F, Berger M, Lam RW, Martiny K, Terman M, Wu JC. Chronotherapeutics (light and wake therapy) in affective disorders. Psychol Med. 2005 Jul;35(7):939-44. doi: 10.1017/s003329170500437x. PMID 16045060
- [Background] Yatham LN, Kennedy SH, O'Donovan C, Parikh S, MacQueen G, McIntyre R, Sharma V, Silverstone P, Alda M, Baruch P, Beaulieu S, Daigneault A, Milev R, Young LT, Ravindran A, Schaffer A, Connolly M, Gorman CP; Canadian Network for Mood and Anxiety Treatments. Canadian Network for Mood and Anxiety Treatments (CANMAT) guidelines for the management of patients with bipolar disorder: consensus and controversies. Bipolar Disord. 2005;7 Suppl 3:5-69. doi: 10.1111/j.1399-5618.2005.00219.x. PMID 15952957
- [Background] Yatham LN, Kennedy SH, O'Donovan C, Parikh SV, MacQueen G, McIntyre RS, Sharma V, Beaulieu S; Guidelines Group, CANMAT. Canadian Network for Mood and Anxiety Treatments (CANMAT) guidelines for the management of patients with bipolar disorder: update 2007. Bipolar Disord. 2006 Dec;8(6):721-39. doi: 10.1111/j.1399-5618.2006.00432.x. PMID 17156158
- [Background] Chaput JP, Despres JP, Bouchard C, Tremblay A. Short sleep duration is associated with reduced leptin levels and increased adiposity: Results from the Quebec family study. Obesity (Silver Spring). 2007 Jan;15(1):253-61. doi: 10.1038/oby.2007.512. PMID 17228054
- [Background] Levitan RD, Masellis M, Basile VS, Lam RW, Kaplan AS, Davis C, Muglia P, Mackenzie B, Tharmalingam S, Kennedy SH, Macciardi F, Kennedy JL. The dopamine-4 receptor gene associated with binge eating and weight gain in women with seasonal affective disorder: an evolutionary perspective. Biol Psychiatry. 2004 Nov 1;56(9):665-9. doi: 10.1016/j.biopsych.2004.08.013. PMID 15522250
- [Background] Krauchi K, Wirz-Justice A, Graw P. High intake of sweets late in the day predicts a rapid and persistent response to light therapy in winter depression. Psychiatry Res. 1993 Feb;46(2):107-17. doi: 10.1016/0165-1781(93)90013-7. PMID 8483971
- [Background] Ortiz-Dominguez A, Hernandez ME, Berlanga C, Gutierrez-Mora D, Moreno J, Heinze G, Pavon L. Immune variations in bipolar disorder: phasic differences. Bipolar Disord. 2007 Sep;9(6):596-602. doi: 10.1111/j.1399-5618.2007.00493.x. PMID 17845274
- [Background] Kupka RW, Breunis MN, Knijff E, Ruwhof C, Nolen WA, Drexhage HA. Immune activation, steroid resistancy and bipolar disorder. Bipolar Disord. 2002;4 Suppl 1:73-4. doi: 10.1034/j.1399-5618.4.s1.29.x. No abstract available. PMID 12479684
- [Background] Lewy AJ, Sack RL, Singer CM, White DM, Hoban TM. Winter depression and the phase-shift hypothesis for bright light's therapeutic effects: history, theory, and experimental evidence. J Biol Rhythms. 1988 Summer;3(2):121-34. doi: 10.1177/074873048800300203. No abstract available. PMID 2979635
- [Background] Lewy AJ, Lefler BJ, Emens JS, Bauer VK. The circadian basis of winter depression. Proc Natl Acad Sci U S A. 2006 May 9;103(19):7414-9. doi: 10.1073/pnas.0602425103. Epub 2006 Apr 28. PMID 16648247
- [Background] Partonen T, Treutlein J, Alpman A, Frank J, Johansson C, Depner M, Aron L, Rietschel M, Wellek S, Soronen P, Paunio T, Koch A, Chen P, Lathrop M, Adolfsson R, Persson ML, Kasper S, Schalling M, Peltonen L, Schumann G. Three circadian clock genes Per2, Arntl, and Npas2 contribute to winter depression. Ann Med. 2007;39(3):229-38. doi: 10.1080/07853890701278795. PMID 17457720
- [Background] O'Brien SM, Scully P, Scott LV, Dinan TG. Cytokine profiles in bipolar affective disorder: focus on acutely ill patients. J Affect Disord. 2006 Feb;90(2-3):263-7. doi: 10.1016/j.jad.2005.11.015. Epub 2006 Jan 10. PMID 16410025